CLINICAL TRIAL: NCT06733974
Title: A Multifaceted Intervention Strategy for Relatives of End-of-life Patients in the Emergency Department: a Cluster Randomized Trial
Brief Title: A Multifaceted Intervention Strategy for Relatives of End-of-life Patients in the Emergency Department
Acronym: MYRIADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP230838; IDRCB no. 2023-A02158-37 (Other: ANSM)
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Grief Disorder, Prolonged
Keywords: Post-traumatic stress disorder (PTSD); prolonged grief disorder (PGD)
MeSH Terms: conditions — Prolonged Grief Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention)
- Multi-faceted Intervention (Experimental)
  Interventions: Other: Multi-faceted Intervention

INTERVENTIONS:
Other: Multi-faceted Intervention — The participant, i.e. relative, will receive the multifaceted intervention which include: a first meeting with the healthcare team including written information about palliative care for dying patients, information on possibility to participate in care, pro-active communication, and dedicated interview and brochure after the patient's death with possibility of psychological follow up.
  Arms: Multi-faceted Intervention

SUMMARY:
In France, a study has reported that about 0.2% of patients visiting the ED died in the ED. A large survey of 145 EDs in 3 French speaking countries has reported that a median of 2 patients dies each week in each ED and its observation unit.

After the death of a loved one, prolonged grief disorder (PGD) is a bereavement-specific syndrome that is defined as intense, prolonged yearning and preoccupation with thoughts of the deceased. PGD prevalence after the loss of a relative was 10% (95%CI 7-14) in the general population.Post-traumatic stress disorder (PTSD) is a mental health condition that is triggered by experiencing a terrifying event. Symptoms may include flashbacks, nightmares, and severe anxiety. The reported lifetime PTSD prevalence is 7% among adults in the general population. Admission and death in the hospital can be a traumatic and stressful experience for relatives, and is associated with an up to 50% risk of PGD and PTSD at 6 months.

In the setting of ICU, several studies have reported that implementation of simple human interventions (information supports including written information on end-of-life care and pro-active communication strategy with systematic interviews with relatives), was associated with a lower risk of PTSD at 3 months (45% vs. 69%) and PGD at 6 months (21% vs 57%). Furthermore, it has been reported that offering the possibility of relatives to be present during nursing and medical care may be beneficial.

In the out of hospital setting, offering the possibility for relative to be present during resuscitation was also associated with a reduction of PTSD at 3 months (15% vs 26%), which was confirmed at 1 year.

The ED setting differs from the one of ICU mainly because exposition time to the dying process is shorter and healthcare workers are less used to manage end of life.

Whether these strategies are beneficial for patients dying in the ED, where dying patients are older with more end- stage chronic diseases and shorter length of stay, remains unknown. The hypothesize of the study is that a multifaceted intervention, including pro-active communication strategy, visual supports, and offering the possibility to be present during nursing and medical care would decrease the risk of PGD in relatives of patients dying in the ED.

ELIGIBILITY:
Inclusion Criteria:

- Relative of a patient, that is dying in the ED, defined by an anticipated life expectancy of less than 72H with previous do not resuscitate order or treatment withholding.

If several relative are present, participation to the trial will be offered in priority to the patient's trustworthy person, the relative most involved in the patient's care, the partner, a parent or child, another family member.

* Age >= 18 years
* Agrees to be followed-up by phone interview at 3 and 6 months
* Informed oral consent
* Relative with health insurance (except AME).

Exclusion Criteria:

* Relative who do not understand, read, or speak French
* Relatives of organ donor patients (these relatives benefit from specific support and communication by the transplant coordination teams)
* Inability to follow up
* Participation in another intervention trial
* Relative under legal protection (tutorship or curatorship)
* Relative deprived of their liberty by a judicial or administrative decision
* Relative physically unable to give his/her oral consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 924 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief 13-item revised scale (PG-R-13) | 6 months after inclusion.
  The PG-R-13 measures the new DSM-V criteria for prolonged grief: yearning, preoccupation, identity disruption, disbelief, avoidance, intense emotional pain, difficulty with reintegration, emotional numbness, feeling that life is meaningless and intense loneliness. The score ranges from 10-50 and a score of 30 or more defined the prolonged grief disorder.

SECONDARY OUTCOMES:
Signs of PTSD assessed by the PCL-5 scale. | 3 months
  20-item self-report measure (about 5-10 min per participan that assesses the 20 DSM-V symptoms of PTSD.
  Each item from 0 ("not at all") to 4 ("extremely) indicate the degree to which they have been bothered by this symptom over the past month. Interpretation of the PCL-5 should be made by a clinician. Scores consist of a total symptom severity score (from 0 to 80) and four subscales:
  * Re-experiencing (items 1-5)
  * Avoidance (items 6-7)
  * Negative alterations in cognition and mood (items 8-14)
  * Hyper-arousal (items 15-20) A cut-off raw score is equal or over 38 for a provisional diagnostic of PTSD.
signs of anxiety and depression HADS scale | 3 months
  This self-assessment scale (about 2-6 min per participant) is divided in two subscores: anxiety subscores (HADS-A) and depression subscores (HADS-D), both containing seven interrelated items. (34) Score for each subscale range from 0 to 21, categorized as follows:
  To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D)
  * Normal < 8
  * Mild to severe equal or over 8

OTHER OUTCOMES:
signs of PTSD | 6 months
  Exploratory outcome: HADS-A and HADS-D respectively assessed by the PCL-5 and HADS scales and any new prescription of antidepressant, anxiolytic, or antipsychotic drugs between inclusion and 6 months.
signs of anxiety | 6 months
  Exploratory outcome: HADS-A and HADS-D respectively assessed by the PCL-5 and HADS scales and any new prescription of antidepressant, anxiolytic, or antipsychotic drugs between inclusion and 6 months.
signs of depression | 6 months
  Exploratory outcome: HADS-A and HADS-D respectively assessed by the PCL-5 and HADS scales and any new prescription of antidepressant, anxiolytic, or antipsychotic drugs between inclusion and 6 months.
satisfaction with communication with the emergency physician and nurse using the medical Interview satisfaction scale (MISS-21) | 3 months after the death
  To assess satisfaction with communication with the emergency physician and nurse, the rapport subscale of the medical interview satisfaction scale (MISS-21) In the intervention group, physicians and nurses complete a questionnaire during the patient's course to evaluate the communication strategy and assess adherence to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency Department Hospital Pitié-Salpêtrière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided